CLINICAL TRIAL: NCT00168727
Title: Zevalin® (Ibritumomab Tiuxetan) Followed by Rituxan® (Rituximab) Maintenance in Previously Treated Low Grade Non-Hodgkin's Lymphoma
Brief Title: Zevalin® Followed by Rituxan® Maintenance in Previously Treated Low Grade Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001-03-ZEV; Former Biogen Idec: 106-I001
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, Low-Grade
Keywords: Radioimmunotherapy; Antigens, CD20
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ibritumomab tiuxetan

INTERVENTIONS:
Drug: ibritumomab tiuxetan (Zevalin®)

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of a treatment regimen using Zevalin® plus Rituxan® for patients who have low grade Non-Hodgkin's Lymphoma (NHL) or relapsed Non-Hodgkin's lymphoma and have been previously treated. This study will use an experimental scheduling regimen. No chemotherapy will be used in this study.

DETAILED DESCRIPTION:
The objective of this study is to determine overall response rate, event-free survival, time-to-progression, time-to-next-therapy, and freedom-from-relapse in patients with low-grade lymphoma in first or second relapse treated with Zevalin followed by 2 years of Rituxan maintenance therapy in a multicenter, community-based setting, as well as evaluate relative response rates in populations with and without prior rituximab therapy, in first versus second relapse, and with and without bulky (> 5 cm in greatest diameter) disease.

To meet the initial trial enrollment goal of 300 patients over two years, 42 total sites were activated. The study has subsequently closed to accrual. Currently 8 sites remain active to follow the 12 subjects enrolled in the past year.

ELIGIBILITY:
Inclusion Criteria:

* Follicular non-Hodgkin's lymphoma including SLL in first or second relapse.
* No anticancer therapy for three wks (six wks if nitrosourea or Mitomycin C); not rituximab refractory.
* Age >= 18 years, not pregnant or lactating.
* Expected survival >= 3 mths; PS 0, 1, or 2.
* ANC >= 1,500/mm3, platelet counts >= 100,000/mm3.
* Total bilirubin > 2.0 mg/dL, creatinine > 2.0 mg/dL.
* Total lymphocyte count < 5,000/mm3 for SLL.
* <25% bone marrow involvement with lymphoma.

Exclusion Criteria:

* Prior ABMT or ASCT, hypocellular or marked reduction in bone marrow precursors, or history of failed stem cell collection.
* Bulky areas of disease more than 10 cm in diameter.
* Patients with CLL, CNS, or mantle cell lymphoma.
* Hx of HIV/AIDS related lymphoma, hepatitis B or C.
* Prior radioimmunotherapy or XRT to >25% of active bone marrow.
* G-CSF or GM-CSF within 2 wks, pegylated G-CSF within 4 wks of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2003-06-01 (Actual); Study Completion 2005-10-31 (Actual)

PRIMARY OUTCOMES:
Determine overall response rate, event-free survival, time-to-progression, time-to-next-therapy, and freedom-from-relapse in pts with low-grade lymphoma in first or second relapse treated with Zevalin® followed by 2 yrs of Rituxan maintenance therapy

SECONDARY OUTCOMES:
Evaluate relative response rates in populations with and without prior rituximab therapy, in first versus second relapse, and with and without bulky (> 5 cm in greatest diameter) disease.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Saville, Study Director — Biogen
Locations (8):
- United States (8):
  - Loma Linda University, Loma Linda, California
  - North County Oncology, Oceanside, California
  - Medical Specialists of Fairfield, Fairfield, Connecticut
  - Queens Hospital, Honolulu, Hawaii
  - Northwest Oncology and Hematology, Elk Grove Village, Illinois
  - Horizon Oncolgy Center, Lafayette, Indiana
  - Specialists in Hematology/Oncology, St Louis, Missouri
  - Presbyterian Hospital Cancer Center, Charlotte, North Carolina